CLINICAL TRIAL: NCT05144516
Title: A Patient-Caregiver Behavioral Intervention for Older Adults With Cancer and Mild Cognitive Impairment-2
Brief Title: Cancer and Mild Cognitive Impairment Dyadic Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00109148
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cancer; Cognitive Impairment
Keywords: Aging; Behavioral Intervention; Mental Health; Communication
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction; Psychological Well-Being; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Caregiver Dyad (Experimental): Participants who are 65 years or older with cancer and mild cognitive impairment with their caregiver.
  Interventions: Behavioral: Behavioral: COPE +

INTERVENTIONS:
Behavioral: Behavioral: COPE + — Six sixty minute sessions that teaches participants distress and communication coping skills.

SUMMARY:
The purpose of this study is to see whether programs that include both a patient and their spouse or a patient and family caregiver (known as a dyad) are helpful for families in which one member of the dyad has cancer and mild memory difficulties and/or concerns. Participant and their spouse or participant and their family caregiver will have six, 60-minute video-conference sessions which will be scheduled at their convenience. The investigator will loan participants a tablet computer (iPad) to use for videoconferencing and train the participant in its use. Participant and their spouse or participant and their family caregiver will complete three assessments - one before starting the sessions, one after the sixth session, and one after 1 month. Each assessment will include surveys, which the participant will complete separately from their spouse or family caregiver. For most people, it will take upwards of 2 - 4 months to complete this study

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria include:

1. Patients with Stage I-IV breast, gastrointestinal (GI), genitourinary (GU), or lung cancer (including extensive stage small cell lung cancer), diagnosed within two years; age 65 or older.
2. Participants must be living at home (either in her/his own home).
3. Participants must be fluent in English and able to learn basic skills for using a tablet computer to conduct videoconference treatment sessions.
4. Exhibit Mild Cognitive Impairment/Concerns
5. Have an informal family caregiver.

Inclusion Criteria:

(Partner or family member) inclusion criteria include:

1. Caregivers are 18 older.
2. Be fluent in English and able to learn basic skills for using a tablet computer to conduct videoconference treatment sessions.
3. Either co-reside with the patient or spend at least 3-4 hours day caregiving.
4. Not exhibit cognitive impairment.

Exclusion Criteria:

1. Participant has visual or hearing impairments that preclude participation.
2. Participant has dementia and do not have the capacity to participate.
3. Have a serious untreated psychiatric illness as documented in medical chart review.
4. The patient and the caregiver score less than a 3 on the National Comprehensive Cancer Network (NCCN) Distress Thermometer (DT) on a scale 0 to 10 to screen for distress. At least one dyad member must experience distress.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of completed sessions as measured by enrollment log | Up to 17 Weeks
Number of participants who are satisfied with the intervention as measured by a score of 24 or greater on the CSQ-8 | Up to 17 weeks
  The Client Satisfaction Questionnaire (CSQ-8) is a self report measure of satisfaction with health and behavioral services received. The CSQ-8 is measured on a four point Likert scale from 1 "Quite Dissatisfied" to 4 "Very Satisfied." Scores range from 8-32, with higher values indicating higher satisfaction

SECONDARY OUTCOMES:
Change in Distress as measured by the DASS-21 | Baseline, up to 17 weeks, up to 1 month follow up
  The Depression, Anxiety, and Stress Scale (DASS-21) measure will be used for rating general distress across three emotional states of depression, anxiety, and stress. The measure has a total of 21 items. Scores range from 0- 63, with higher scores indicating greater distress.
Change in Quality of Life as measured by the FACT-G | Baseline, up to 17 weeks, up to 1 month follow up
  The Functional Assessment of Cancer Therapy: General (FACT-G) measure will be used for rating quality of life. The measure has a total of 27 items. Scores range from 0-108, with higher scores indicating greater quality of life.
Change in Communication Patterns as measured by the CPQ-SF | Baseline, up to 17 weeks, up to 1 month follow up
  The Communication Patterns Questionnaire Short-Form (CPQ-SF) will be used for rating communication patterns in a relationship. The measure has a total of 11 items. Scores range from 11-99, higher scores indicate a greater likelihood of using a particular communication pattern during conflict interactions.
Change in Relationship Satisfaction as measured by the Mutuality Scale of the Family Care Inventory | Baseline, up to 17 weeks, up to 1 month follow up
  The Mutuality Scale of the Family Care Inventory will be used for rating mutual concerns and overall relationship satisfaction. The measure consists of 15 items. Scores range from 0-60, higher scores indicate greater relationship satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ramos, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No